CLINICAL TRIAL: NCT04671030
Title: Effects of the Addition of a Prokinetic Agent to Thrice Weekly Bowel Care in Individuals With SCI
Brief Title: Use of a Prokinetic Agent as an Adjunct to Thrice Weekly Bowel Care After SCI
Acronym: TWBC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Mark Korsten, Chief of Gastroenterology, James J. Peters Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KOR-12-35
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Spinal Cord Injuries; Constipation; Neurogenic Bowel
Keywords: Neostigmine; Glycopyrrolate; Transdermal; Intravenous; Constipation; Bowel care; Neurogenic bowel
MeSH Terms: conditions — Spinal Cord Injuries; Constipation; Neurogenic Bowel | interventions — Neostigmine; Glycopyrrolate; Iontophoresis

STUDY DESIGN:
Intervention Model Description: Single group interventional study with brief crossover of subjects into the placebo group
Who Masked: Participant
Masking Description: Subjects are not aware of the nature of the drug that they are receiving
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Treatment group (Experimental): Subjects are screened by criteria, intravenous and transdermal iontophoresis then undergo the study during which they will be administered the placebo alternating with real drug without being aware of which is being given.
  Interventions: Drug: Neostigmine and Glycopyrrolate; Device: Iontophoresis
- Placebo group (Placebo Comparator): Placebo will be given without the subject being aware of the time in advance.
  Interventions: Device: Iontophoresis

INTERVENTIONS:
Drug: Neostigmine and Glycopyrrolate — Intravenous followed by transdermal administration of the two drug combination.
  Arms: Treatment group
Device: Iontophoresis — Application of direct current to skin using an FDA-approved device
  Other Names: I-Box

SUMMARY:
To measure a baseline for each subject, an abdominal x-ray (KUB) was performed, the SCI Bowel Survey and Treatment Satisfaction Questionnaire (TSQM) were administered and the subject's weight determined. After all the baseline measurements were acquired, the subjects underwent transdermal screening with hair epilation to test their response to transdermal administration of NEO (0.07mg/kg) and GLY (0.014mg/kg). All subjects had a positive response (bowel movement within 60 minutes of drug administration) and received five more cycles of bowel care for two weeks. All subjects reported bowel evacuation during each session and some reported side effects like slight dry mouth, eye twitching, and cramping. These side effects lasted approximately 20-30 minutes in duration and there were no clinically significant changes in cardiopulmonary vital signs. Six subjects after completing two weeks of bowel care had an abdominal x-ray (KUB) done. Also, they were weighted and reassessed using the TSQM and bowel survey.

DETAILED DESCRIPTION:
Part 1: IV Screening Twenty subjects with chronic SCI (>1 year) and difficulty with evacuation (DWE) managed by a regular, thrice weekly bowel care (BC) routines will be recruited for study participation. In order to determine eligibility for the study, the subject will have to undergo an IV screening to test whether or not they are responsive to the drug treatment (neostigmine-glycopyrrolate). Subjects will receive the following dose: 0.03mg/kg neostigmine (NEO) and 0.006mg/kg glycopyrrolate (GLY). If the subject responds (bowel movement) to the IV treatment, they will be allowed to continue on to part 2 of the study. If patient does not have a successful bowel movement, then they will be considered a non-responder and study participation will be discontinued. Study procedures can be found in table below.

Part 2: Baseline and Iontophoresis Screening Once eligibility has been determined, and subject consent has been obtained, each subject will undergo 1 week of baseline observation. An abdominal x-ray (KUB) will be performed, the SCI Bowel Survey and Treatment Satisfaction Questionnaire (TSQM) will be administered, and the subject's weight determined. Each subject will continue with regular bowel care and after 1 week, all of the baseline measurements (KUB, weight and surveys) will be repeated. This will be followed by an additional screening visit during which we will concomitantly administer transcutaneous NEO and GLY via iontophoresis (ION). Subjects will receive the following dose: 0.07mg/kg NEO and 0.014mg/kg GLY. This visit will be scheduled on a BC day. All procedures will take place in the "Blue Room" located in the SCI ward. As part of the setup, subjects will be instrumented with blood pressure cuff; intravenous access will be obtained at a peripheral vein (if one is not available), as a precautionary measure, since the drug will be administered via an Iontophoresis transdermal patch. Heart rate will be continuously monitored throughout the procedure through finger oximetry. Symptoms will be assessed every 5 minutes for 60 minutes. Impulse Oscillometry system (IOS) will be used to measure the effect of the medication on airway obstruction. If the subject has a positive response (bowel movement within 60 minutes of drug administration) he/she will be eligible to continue to the third study phase. If the subject does not respond, the subject will be considered a non-responder and study participation will be discontinued. We expect that about 1/3rd of the subjects will be non-responders, or will be lost to attrition; therefore, we are prepared to over-recruit by 5 subjects in order to ensure that at least 15 subjects will be eligible to complete the second part of the study.

The study will be stopped once the patient experiences a bowel movement within 30 minutes of administering ION NEO because the protocol objective will have been achieved. If the patient should experience cardiopulmonary side effects when receiving the ION NEO that are not effectively reversed by the ION GLY, the study will be stopped. In addition, the study investigators reserve the right to stop the study should they have any other safety concerns.

Part 3: 2 Week Treatment Each subject will be assessed for their perception of their current BC routine using the Treatment Satisfaction Questionnaire for Medication (TSQM-Appendix 1), and their bowel habits using the bowel survey (Appendix 2).The subject will then be asked to continue with their normal BC routine for two weeks, with the exception that NEO and GLY will be administered at the beginning of each BC session as an adjunct to each subject's normal routine. Subjects will be asked to come to the JJPVAMC for each BC session. Each BC session will be documented by a study team member including the time needed to complete BC, methods used (i.e. number of enemas used, oral laxatives, suppositories, digital stimulation, abdominal massage) and the quality and completeness of the bowel movement. Heart rate, oxygenation and blood pressure will be monitored continuously. Subjects will be weighed at baseline, once after each week of treatment and once at the post treatment follow-up visit. After two weeks of treatment, each subject will undergo a final KUB and be reassessed for their perception of the BC routine for the past two weeks using the TSQM and their bowel habits (bowel survey).

*During the treatment period (part 3), monitoring will take place for the first hour after administration of study medications. However, bowel care will continue for as long as is clinically indicated. Additional techniques for bowel care (i.e. enema, suppository, digital stimulation, etc.) will be used in coordination with SCI nurses to promote bowel evacuation for subjects who do not respond.

**An IV line will be inserted during all study visits. Study medication will be administered intravenously during Part 1 only. An IV line will be available however through all sessions involving study medication for safety purposes in the case that an antidote needs to be administered

ELIGIBILITY:
1. Inclusion Criteria:

   * Spinal Cord Injury:
   * Level of injury C1 to S4
   * Duration of injury over 1 year
   * Excess time for bowel evacuation (over 60 minutes per bowel training session).
2. Exclusion Criteria:

   * Previous Adverse Reaction or Hypersensitivity to Electrical Stimulation
   * Do not require additional bowel care or have "normal bowel function"
   * Known sensitivity to Neostigmine and Glycopyrrolate
   * Blockage in Bowel or Bladder
   * Myocardial Infarction in the past 6months
   * Blood Pressure over 160 over 100 mg Hg with being on 3 or more different classes of antihypertensive medications
   * Organ Damage (heart and kidney) and/or TIA, CVA as a result of hypertension
   * Known past history of coronary artery disease, chronic heart failure, bradyarrythmia
   * Slow Heart Rate (under 45 bpm)
   * Active respiratory diseases
   * Known history of asthma during lifetime
   * Recent (within 3 months) respiratory infections
   * Adrenal Insufficiency
   * Pregnancy or potential for pregnancy
   * Lactating/nursing females
   * Use of any antibiotics in past 7 days
   * Use of medications known to affect respiratory system
   * Concurrent participation in other clinical trials (within 30 days)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Time to first bowel evacuation | within 1 hour
  Measured from completion of adminstration to first bowel evacuation

CONTACTS AND LOCATIONS:
Locations (1):
- James J Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No